CLINICAL TRIAL: NCT01598116
Title: A Prospective Longitudinal Study to Identify Biomarkers in Children With Hemangiomas.
Status: Completed | Type: Observational
Sponsor: Gayle Gordillo (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 10-00482
Record Dates: First submitted 2012-01-13; First posted 2012-05-15 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Urine Specimen Collection; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemangioma: Identify biomarkers in children with hemangiomas.
  Interventions: Procedure: Urine collection and ultrasonography
- Without Hemangioma: Age-matched controlled group without hemangioma.
  Interventions: Procedure: Urine collection

INTERVENTIONS:
Procedure: Urine collection and ultrasonography — Bagged urine collection and ultrasound at each visit
  Groups: Hemangioma
Procedure: Urine collection — Bagged urine collection
  Groups: Without Hemangioma

SUMMARY:
Current treatment options for hemangiomas, such as propranolol, steroids and interferon, all have the potential for significantly harmful side effects. The purpose of this study is to identify potential biomarkers that can be used to design clinical trials and accelerate the delivery of new treatment alternatives to children with hemangiomas.

DETAILED DESCRIPTION:
Urine will be collected from children with hemangiomas and age-matched healthy controls at 2,4,6,9,12,18 and 24 months of age. Children with hemangiomas will also have ultrasound examination performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Children with hemangioma
* Age ≤ 5 months
* Doppler ultrasound confirmed diagnosis of hemangioma to rule out presence of vascular malformation
* Age matched control ≤ 5 months (no hemangioma)

Exclusion Criteria:

* Hemangioma treated prior to or during study period with laser, steroids, interferon, or propranolol, or any other drug or device intended to inhibit the growth of the hemangioma
* Known history of sickle cell anemia, thalassemia, or other hemoglobinopathy
* Hemangioma presented as fully formed at birth consistent with rapidly involuting or non-involuting congenital hemangioma
* PHACES syndrome- posterior fossa malformations, hemangioma, arterial anomalies, cardiac anomalies, eye abnormalities, sternal anomalies
* Parent/guardian unable to speak english to provide informed consent and no interpreter is present

Ages: 4 Weeks to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with hemangiomas and children without hemangiomas will be enrolled from Hemangioma and Vascular Malformation Clinic and Ambulatory Pediatric Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-12-12 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Chemically modified DNA | 6 months
  Determine whether changes in urinary 8-OHdG can be used as biomarkers for HE growth and involution.

SECONDARY OUTCOMES:
Blood flow velocity | 6 months
  Obtain Doppler ultrasound measurements of HE blood flow velocity and size on the same days as serum and urine specimen collection to determine whether changes in blood flow velocity and size correlate with changes in 8-OHdG production.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M Gordillo, MD, Principal Investigator — Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States